CLINICAL TRIAL: NCT04429048
Title: Effect of Acupressure at PC6 on Headache in Patients With Migraine: Single-blinded, Randomized, Controlled Clinical Trial
Brief Title: Effect of Acupressure in Migraine: Single-blinded, Randomized, Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202002094RIND
Record Dates: First submitted 2020-05-24; First posted 2020-06-11 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Migraine; Status
Keywords: migraine ,acupressure,CGRP,neurokinin A
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure group (Experimental): The participants received modern routing standard therapy accompanied with the round plastic studs of sea-band were placed just on the skin surface of bilateral PC6 acupoints , and then keep the persistent compressive state for 3 minutes per time and three times a day.
  Interventions: Device: Acupressure elastic band (Sea-Band)
- control group (Sham Comparator): The participants received modern routing standard therapy only with general elastic band without bud over PC6 acupoints.
  Interventions: Device: General elastic band (no bud)

INTERVENTIONS:
Device: Acupressure elastic band (Sea-Band) — The PC6 acupressure was done via Sea-Band in persistent compressive state for 3 minutes per time and three times a day , then at least 5 days in one week for 6 weeks continuously except modern routine standard therapy
  Arms: acupressure group
Device: General elastic band (no bud) — general elastic band was put over bilateral PC6 acupoints
  Arms: control group

SUMMARY:
Background :

Migraine is one of the most complex, prevalent, debilitating neurologic disorder in the world. In clinical experience, there are limitation over western medicine for migraine, especially some extra adverse effects. In traditional Chinese medicine(TCM), there are some reviews and clinical practice point out acupressure at PC6 could relieve nausea/ vomiting and pain while migraine. Recent researches also mention Calcitonin gene-related peptide (CGRP) and Neurokinin A (NKA) in some degree correlated with the mechanism of migraine.

Objective:

CGRP and NKA play vital roles of migraine. In comparison with oral medication only and PC6 acupressure via oral medication, if there were better effect for migraine control. In addition, investigators evaluate the plasma CGRP and NKA level before and after study to figure out if any positive value and any correlation with acupressure.

Method:

By single-blinded, randomized, controlled clinical trial, total of 56 patients with migraine were divided equally into acupressure group (modern routing standard therapy plus PC6 acupressure) and control group (modern routing standard therapy). Before intervention, the participants needed to finish the Migraine Disability Assessment (MIDAS) questionnaire evaluation. After 6 weeks, investigators will evaluate the severity, frequencies of headaches and pain-killer consumption as primary outcome. In addition, investigators will investigate if there were change of serum CGRP/NKA level after 6 weeks and the score changes of MOS 36-Item Short-Form Health Survey as secondary outcome.

Expected results:

The investigators predict that PC6 acupressure may not only reduce severity, frequencies and duration of headaches but also reduce the dose of NSAIDs. In addition, the PC6 acupressure also may reduce levels of serum CGRP and NKA, and improve the quality of life meanwhile.

DETAILED DESCRIPTION:
Introduction:

Migraine is one of the most complex, prevalent, debilitating neurologic disorder and the prevalence higher in female group. In general, there are many kinds of therapy for migraine nowadays including of acute abortion oral drugs such as triptan, ergotamine, non-steroid anti-inflammatory drugs, acetaminophen and preventive agents such as calcium channel blocker (Flunarizine), anti-epileptic drugs (valproic acid, Topiramate, Pregabalin), beta adrenergic-blocker (Propranolol), Selective Serotonin Reuptake Inhibitors(SSRI), anti-emetic agents (Prochlorperazine) and other injection therapy such as Onabotulinum Toxin A or CGRP (Calcitonin gene-related peptide) antagonist etc. The CGRP plays an important role of trigemino-vascular responses in migraine. The serum CGRP levels elevated while migraine attack and chronic migraine, therefore, CGRP is a potential biomarker. In recent studies, higher plasma CGRP level during interictal phase of migraine or chronic migraine is indicated the better response for Onabotulinum Toxin A and reduced plasma CGRP level can relieve the discomfort of migraine. Neurokinin A (NKA) levels of venous blood are significantly higher in responders than these nonresponse before the rizatriptan treatment, whereas reduced the levels of both CGRP and NKA one hours after the treatment . The headache is associated with nausea in about 80% of episodes, vomiting in about 30% in patients with migraine.

PC6 is belong to pericardium meridian locates the anterior aspect of forearm between the tendons of the palmaris longus and the flexor carpi radialis, 2 cun proximal to the wrist transverse stripes just on the median nerve . The antiemetic is lower for preventing postoperative nausea and vomiting in the combination PC6 acupoint stimulation than these patients with antiemetic only. Acupuncture at the PC6 is an effective alternative treatment to conventional pharmacological treatment and resulted in almost immediate cessation of intraoperative nausea and vomiting. Therefore, acupressure at PC6 is an effective and safety method for nausea and vomiting. In addition, stimulation at PC6 can activate hypothalamic orexin neurons, and that release orexins to induce analgesia. Taken together, PC6 stimulation can produce effect of both analgesia and antiemetic effects. The present study suppose stimulation at PC6 is beneficial for the treatment of migraine.

Therefore, the investigators designed a single-blinded, randomized, controlled trial to evaluate the effect of acupressure at PC6 on headache in patients with migraine.

Method and study design:

(A) Participants The patients with migraine were enrolled from the outdoor patients (OPD) of neurological department, Yunlin branch of National Taiwan University hospital. The basic laboratory data including peripheral blood cells, Na/K/Ca/Mg, alanine aminotransferase (ALT), creatinine, iron/total iron-binding capacity (TIBC)/ferritin to exclude extremely abnormal metabolic disturbance or liver/renal functional impairment which may cause secondary headache; and the awake electroencephalography (EEG) and brain image including computer tomography (C-T) or magnetic resonance image (MRI) also were done to rule out any intracranial structure lesion prior to the trial.

The migraine was diagnosed according to clinical manifestation and criteria from beta version of the third edition of the International Classification of Headache Disorders (ICHD-3). In addition, non-steroid anti-inflammatory drugs (NSAIDs) are used as episodic way while migraine attack and Propranolol (Inderal R) is used as preventive way no matter when migraine attack. In addition, the participants needed to finish the Migraine Disability Assessment (MIDAS) questionnaire evaluation of 6 weeks.

(B) Study design: Single-blinded, randomized, controlled clinical trial. (C) Assessment time: before PC6 acupressure (V1), two weeks after acupressure (V2), four weeks after acupressure (V3) and six weeks after acupressure (D) Statistical analysis : Categorical data will be displayed in numbers and percentages, whereas continuous variables will be given as means ± standard deviations or median (Q1, Q3). Differences in categorical variables will be tested using the chi-square test or Fisher exact test and differences in continuous variables will be tested using the two sample independent t test or Mann-Whitney test between groups. The generalized estimating equations (GEE) will be used to compare the change of primary outcomes over time (the four time points (V1-V4)) between two groups. A p value of less than 0.05 will be considered statistically significant. All statistical analyses will be performed using SPSS Statistics 24or R version 3.4.4 .

Outcome :

The study of the present study predicts that PC6 acupressure may reduce severity of headaches, the frequency of headache attacks and duration of headache, and also reduce the dose of NSAID. In addition, the PC6 acupressure also may reduce levels of serum CGRP and NKA, and also may improve the quality of life.

ELIGIBILITY:
A. Inclusion criteria

1. Age ranged from 20 to 50-year-old (inclusion)
2. Female or male.
3. Neurological examination was within normal limit.
4. Neither epileptiform discharge from EEG nor abnormality of neuroimage

B. Exclusion criteria

1. Headache was results from adverse effects for NSAIDs and Propranolol.
2. Active skin lesion or oozing wound over PC6 acupoints.
3. Pregnancy or lactation.
4. Recent traumatic brain injury or brain tumor.
5. Secondary headache
6. Brain surgical history.
7. Refuse sign informed consent.
8. Extremely abnormal metabolic disturbance (such as iron deficiency anemia, hypo/hypernatremia, hypo/hyperkalemia, hypo/hypercalcemia, hypo/ hypermagnesemia) and liver/renal dysfunction ALT > 3x normal upper limits; creatinine >1.4)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Headache duration | After 6 weeks , evaluate how many episodes of lesser duration(<4hours) of the two groups
  duration (if attack less than 4hours which means better response)
Headache severity | After 6 weeks, evaluate the headache severity (VAS score) if any decreased
  Severity by visual analog scale (0~10), if VAS score decreased 2 points which means better results
Headache frequency | evaluate total headache episodes after 6 weeks
  how many times headache occurred (if attack < 8 times which means effective)
dosage of pain killers | evaluation total amount of pain-killer consumption after 6 weeks
  how many dosage of pain kill taken (if pain killer taken less than 20 pills which means effective therapy)

SECONDARY OUTCOMES:
Calcitonin gene-related peptide (CGRP) level | 1st time: 1 day of sign informed consent ; 2nd time: through study completion, an average of 6 weeks
  Check serum CGRP level to evaluate the correlation
Neurokinin A (NKA) level | 1st time: 1 day of sign informed consent ; 2nd time: through study completion, an average of 6 weeks
  Check NKA level to realize any discrepancy
the score of 36-Item Short Form Health Survey (SF-36) | through study completion, an average of 6 weeks
  Complete form for quality evaluation (score: 0~100, worse to better)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-hung Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin County, Taiwan